CLINICAL TRIAL: NCT05058404
Title: Shortened vs Standard Chemotherapy Combined With Immunotherapy for the Initial Treatment of Patients With High Tumor Burden Follicular Lymphoma. A Randomized, Open Label, Phase III Study by Fondazione Italiana Linfomi.
Brief Title: Shortened vs Standard Chemotherapy Combined With Immunotherapy for the Initial Treatment of Patients With High Tumor Burden Follicular Lymphoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIL_FOLL19
Record Dates: First submitted 2021-09-07; First posted 2021-09-27 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-06

CONDITIONS: Follicular Lymphoma
Keywords: High tumor burden Follicular Lymphoma; Shortened vs standard chemotherapy; Immunotherapy; Initial treatment
MeSH Terms: conditions — Lymphoma, Follicular | interventions — R-CHOP protocol

STUDY DESIGN:
Intervention Model Description: This is a prospective, multicenter, phase III, two arms randomized trial with a non-inferiority design with Progression-Free Survival (PFS) as primary endpoint. Patients who meet all eligibility criteria will be centrally randomized to one of the two treatment arms in a 1:1 ratio, using random sequences blocks of variable size. The web-based allocation process, completely concealed to researchers, will be stratified according Follicular Lymphoma International Prognostic Index 2 (FLIPI2) score (0-2, 3-5), chemotherapy regimen (CHOP, Bendamustine, CVP) and anti-CD20 Monoclonal Antibody (MoAb) (rituximab, obinutuzumab). A non-inferiority design has been adopted to demonstrate that a shortened exposure to chemotherapy in patients responding to the first four cycles of immunochemotherapy is not detrimental in terms of PFS compared to full dose standard treatment. The primary comparison will be done as an Intention To Treat (ITT) analysis including all randomized patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard arm (A) (Experimental): Patients will start immunochemotherapy with one of the approved regimens (R-CHOP, R-Bendamustine, G-CHOP, G-Bendamustine, G-CVP).
  Patients randomized to Arm A will receive an induction immunochemotherapy at full doses (standard schedule).
  After cycle 4, patients will be assessed for response and will complete their planned therapy if at least a stable disease is confirmed.
  At the end of induction responding patients (CR, PR) will be addressed to a standard anti-CD20 maintenance (1 dose every 8 weeks for two years) with the same Monoclonal Antibody (MoAb) given during induction.
  Interventions: Drug: Immunochemotherapy regimen: Rituximab-bendamustine (Arm A); Drug: Immunochemotherapy regimen: R-CHOP (Arm A); Drug: Immunochemotherapy regimen: G-bendamustine (Arm A); Drug: Immunochemotherapy regimen: G-CHOP (Arm A); Drug: Immunochemotherapy regimen: G-CVP (Arm A)
- Experimental arm (B) (Experimental): Patients will start immunochemotherapy with one of the approved regimens (R-CHOP, R-Bendamustine, G-CHOP, G-Bendamustine, G-CVP).
  Patients randomized to Arm B will start their induction treatment with 4 cycles of the immunochemotherapy standard dose chosen by the physician: after cycle 4, patients will be assessed for response and will proceed with subsequent treatment based on the quality of their response. Specifically:
  * Patients achieving a CR will receive a shortened treatment: in detail, they won't receive any further chemotherapy but will complete induction with 4 additional cycles of only the Monoclonal Antibody (MoAb) given during the first four cycles;
  * In case if response less than CR, (PR,SD), patients will complete treatment as planned for patients in Arm A.
  At the end of induction responding patients (CR, PR) will be addressed to a standard anti-CD20 maintenance (1 dose every 8 weeks for two years) with the same Monoclonal Antibody (MoAb) given during induction.
  Interventions: Drug: Immunochemotherapy regimen: Rituximab-bendamustine (Arm B); Drug: Immunochemotherapy regimen: R-CHOP (Arm B); Drug: Immunochemotherapy regimen: G-bendamustine (Arm B); Drug: Immunochemotherapy regimen: G-CHOP (Arm B); Drug: Immunochemotherapy regimen: G-CVP (Arm B)

INTERVENTIONS:
Drug: Immunochemotherapy regimen: Rituximab-bendamustine (Arm A) — Arm A (Standard arm):
  4 cycles of Rituximab-bendamustine Q28 (28-days cycles); Patients will undergo an early restaging after cycle 4: those with at least a stable disease will complete the induction treatment with 2 cycles of R-bendamustine Q28 + 2 cycles Q28 of rituximab;
  Both Arms:
  Whichever the regimen, in responding patients (Complete Remission CR, Partial Remission PR) at the end of induction a standard maintenance will follows (1 dose every 8 weeks for 2 years) with the same anti-CD20 Monoclonal Antibody (MoAb) used for induction.
  Patients in both arms with progressive disease at any time and patients in stable disease (SD) at the End Of Induction (EOI) shall be considered for salvage therapy at clinician discretion.
  Other Names: R-Benda, R-bendamustine
  Arms: Standard arm (A)
Drug: Immunochemotherapy regimen: Rituximab-bendamustine (Arm B) — Arm B (Experimental arm):
  4 cycles of Rituximab-bendamustine Q28 (28-days cycles);
  After cycle 4 patients will undergo an early restaging. Induction therapy shall be completed based on the response achieved and on the treatment chosen as below specified:
  * if in CR: patients will receive no more chemotherapy but will complete induction with the MoAb only, in this case: 4 cycles of rituximab;
  * if less than CR (PR, SD): the immunochemotherapy program will be completed as outlined for Arm A: 2 cycles of R-bendamustine Q28 + 2 cycles Q28 of rituximab;
  Both Arms:
  Whichever the regimen, in responding patients (CR, PR) at the end of induction a standard maintenance will follows (1 dose every 8 weeks for 2 years) with the same anti-CD20 Monoclonal Antibody (MoAb) used for induction.
  Patients in both arms with progressive disease at any time and patients in SD at the End Of Induction (EOI) shall be considered for salvage therapy at clinician discretion.
  Other Names: R-Benda, R-bendamustine
  Arms: Experimental arm (B)
Drug: Immunochemotherapy regimen: R-CHOP (Arm A) — Arm A (Standard arm):
  4 cycles of R-CHOP Q21 (21-days cycles); R-CHOP = Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, Prednisone
  Patients will undergo an early restaging after cycle 4: those with at least a stable disease will complete the induction treatment with 2 cycles of R-CHOP Q21 + 2 cycles Q21 of rituximab;
  Both Arms:
  Whichever the regimen, in responding patients (Complete Remission CR, Partial Remission PR) at the end of induction a standard maintenance will follows (1 dose every 8 weeks for 2 years) with the same anti-CD20 Monoclonal Antibody (MoAb) used for induction.
  Patients in both arms with progressive disease at any time and patients in stable disease (SD) at the End Of Induction (EOI) shall be considered for salvage therapy at clinician discretion: these patients will be included in the analysis planned by the study.
  Other Names: R-CHOP
  Arms: Standard arm (A)
Drug: Immunochemotherapy regimen: R-CHOP (Arm B) — Arm B (Experimental arm):
  4 cycles of R-CHOP Q21 (21-days cycles); R-CHOP = Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, Prednisone
  After cycle 4 patients will undergo an early restaging: induction therapy shall be completed based on the response achieved and on the treatment chosen:
  * if in CR: patients will receive no more chemotherapy but will complete induction with the MoAb only, in this case: 4 cycles of rituximab;
  * if less than CR (PR, SD): the immunochemotherapy program will be completed as outlined for Arm A: 2 cycles of R-CHOP Q21+ 2 cycles Q21of rituximab
  Both Arms: in responding patients (CR, PR) at the end of induction a standard maintenance will follows (1 dose every 8 weeks for 2 years) with the same anti-CD20 MoAb used for induction.
  Patients in both arms with progressive disease at any time and patients in SD at the EOI shall be considered for salvage therapy at clinician discretion: these patients will be included in the analysis.
  Other Names: R-CHOP
  Arms: Experimental arm (B)
Drug: Immunochemotherapy regimen: G-bendamustine (Arm A) — Arm A (Standard arm):
  4 cycles of G-bendamustine Q28 (28-days cycles); G-Bendamustine = Obinutuzumab and Bendamustine
  Patients will undergo an early restaging after cycle 4: those with at least a stable disease will complete the induction treatment with 2 cycles of G-bendamustine Q28 (28-days cycles);
  Both Arms:
  Whichever the regimen, in responding patients (Complete Remission CR, Partial Remission) at the end of induction a standard maintenance will follows (1 dose every 8 weeks for 2 years) with the same anti-CD20 Monoclonal Antibody (MoAb) used for induction.
  Patients in both arms with progressive disease at any time and patients in Stable Disease SD at the End Of Induction (EOI) shall be considered for salvage therapy at clinician discretion.
  Other Names: G-Benda
  Arms: Standard arm (A)
Drug: Immunochemotherapy regimen: G-bendamustine (Arm B) — Arm B (Experimental arm):
  4 cycles of G-bendamustine Q28 (28-days cycles); G-Bendamustine = Obinutuzumab and Bendamustine
  After cycle 4 patients will undergo an early restaging. Induction therapy shall be completed based on the response achieved and on the treatment chosen as below specified:
  * if in CR: patients will receive no more chemotherapy but will complete induction with the Monoclonal Antibody (MoAb) only, in this case 2 cycles of obinutuzumab;
  * if less than CR (PR, SD): the immunochemotherapy program will be completed as outlined for Arm A: 2 cycles of G-bendamustine Q28;
  Both Arms: in responding patients (CR, PR) at the end of induction a standard maintenance will follows (1 dose every 8 weeks for 2 years) with the same anti-CD20 (MoAb) used for induction.
  Patients in both arms with progressive disease at any time and patients in SD at the End Of Induction (EOI) shall be considered for salvage therapy at clinician discretion.
  Other Names: G-Benda
  Arms: Experimental arm (B)
Drug: Immunochemotherapy regimen: G-CHOP (Arm A) — Arm A (Standard arm):
  4 cycles of G-CHOP Q21 (21-days cycles) G-CHOP = Obinutuzumab, Cyclophosphamide, Doxorubicin, Vincristine, Prednisone
  Patients will undergo an early restaging after cycle 4: those with at least a stable disease will complete the induction treatment with 2 cycles of G-CHOP Q21 + 2 cycles Q21 of obinutuzumab;
  Both Arms:
  Whichever the regimen, in responding patients (Complete Remission CR, Partial Remission PR) at the end of induction a standard maintenance will follows (1 dose every 8 weeks for 2 years) with the same anti-CD20 Monoclonal Antibody (MoAb) used for induction.
  Patients in both arms with progressive disease at any time and patients in stable disease (SD) at the End Of Induction (EOI) shall be considered for salvage therapy at clinician discretion.
  Other Names: G-CHOP
  Arms: Standard arm (A)
Drug: Immunochemotherapy regimen: G-CHOP (Arm B) — 4 cycles of G-CHOP Q21 (21-days cycles) G-CHOP = Obinutuzumab, Cyclophosphamide, Doxorubicin, Vincristine, Prednisone
  After cycle 4 patients will undergo an early restaging. Induction therapy shall be completed based on the response achieved and on the treatment chosen as below specified:
  * if in CR: patients will receive no more chemotherapy but will complete induction with the Monoclonal Antibody (MoAb) only, in this case: 4 cycles of obinutuzumab;
  * if less than CR (PR, SD): the immunochemotherapy program will be completed as outlined for Arm A: 2 cycles of G-CHOP Q21 + 2 cycles Q21 of obinutuzumab;
  Both Arms: in responding patients (CR, PR) at the end of induction a standard maintenance will follows (1 dose every 8 weeks for 2 years) with the same anti-CD20 MoAb used for induction.
  Patients in both arms with progressive disease at any time and patients in SD at the EOI shall be considered for salvage therapy at clinician discretion.
  Other Names: G-CHOP
  Arms: Experimental arm (B)
Drug: Immunochemotherapy regimen: G-CVP (Arm A) — Arm A (Standard arm):
  4 cycles of G-CVP Q21 (21-days cycles) G-CVP = Obinutuzumab, Cyclophosphamide, Vincristine, Prednisone.
  Patients will undergo an early restaging after cycle 4: those with at least a stable disease will complete the induction treatment with 4 cycles of G-CVP Q21;
  Both Arms:
  Whichever the regimen, in responding patients (Complete Remission CR, Partial Remission PR) at the end of induction a standard maintenance will follows (1 dose every 8 weeks for 2 years) with the same anti-CD20 Monoclonal Antibody (MoAb) used for induction.
  Patients in both arms with progressive disease at any time and patients in stable disease SD at the End Of Induction (EOI) shall be considered for salvage therapy at clinician discretion.
  Other Names: G-CVP
  Arms: Standard arm (A)
Drug: Immunochemotherapy regimen: G-CVP (Arm B) — Arm B (Experimental arm):
  4 cycles of G-CVP Q21 (21-days cycles) G-CVP = Obinutuzumab, Cyclophosphamide, Vincristine, Prednisone.
  After cycle 4 patients will undergo an early restaging. Induction therapy shall be completed based on the response achieved and on the treatment chosen as below specified:
  * if in CR: patients will receive no more chemotherapy but will complete induction with the Monoclonal Antibody (MoAb) only, in this case: 4 cycles of obinutuzumab;
  * if less than CR (PR, SD): the immunochemotherapy program will be completed as outlined for Arm A: 4 cycles of G-CVP Q21
  Both Arms: in responding patients (CR, PR) at the end of induction a standard maintenance will follows (1 dose every 8 weeks for 2 years) with the same anti-CD20 MoAb used for induction.
  Patients in both arms with progressive disease at any time and patients in SD at the End Of Induction (EOI) shall be considered for salvage therapy at clinician discretion.
  Other Names: G-CVP
  Arms: Experimental arm (B)

SUMMARY:
FIL_FOLL19 is an open-label, multicenter, randomized phase III trial. The sponsor of this clinical trial is Fondazione Italiana Linfomi (FIL).

The Primary Objective of the study is to demonstrate that, in patients with newly diagnosed, advanced stage Follicular Lymphoma (FL) with high tumor burden according to the Groupe d'Etude des Lymphomes Folliculaires (GELF) criteria, a treatment strategy that reduces the number of chemotherapy cycles in case of early response to immunochemotherapy is not inferior compared to standard therapy at full dose in terms of Progression-Free Survival (PFS).

DETAILED DESCRIPTION:
This is an open-label, multicenter, randomized phase III trial. The study plans to randomize patients with a 1:1 ratio to Arm A (Standard arm) or Arm B (Experimental arm).

Once randomized, each patient will start immunochemotherapy with one of the approved regimens (R-CHOP, R-Bendamustine, G-CHOP, G-Bendamustine, G-CVP) chosen by the physician on a patient basis before randomization.

Patients randomized to Arm A will receive an induction immunochemotherapy at full doses (standard schedule).

After cycle 4, patients will be assessed for response and will complete their planned therapy if at least a stable disease is confirmed.

Patients randomized to Arm B will start their induction treatment with 4 cycles of the immunochemotherapy standard dose chosen by the physician: after cycle 4, patients will be assessed for response and will proceed with subsequent treatment based on the quality of their response.

Specifically:

* Patients achieving a Complete Remission (CR) will receive a shortened treatment: in detail, they won't receive any further chemotherapy but will complete induction with 4 additional cycles of only the Monoclonal Antibody (MoAb) given during the first four cycles (in case of G-bendamustine, 2 additional cycles of obinutuzumab);
* In case if response less than Complete Remission (CR), Partial Remission (PR) or Stable Disease (SD), patients will complete treatment as planned for patients in Arm A.

In both arms, at the end of induction responding patients (CR, PR) will be addressed to a standard anti-CD20 maintenance (1 dose every 8 weeks for two years) with the same Monoclonal Antibody (MoAb) given during induction.

Patients with progressive disease at any time (regardless of treatment arm) will be addressed to salvage therapy.

The study plans the evaluation of quality of life by collecting the Patient-Reported Outcome(s) (PROs) through the Functional Assessment of Cancer Treatment-Lymphoma (FACT-Lym questionnaire) at predetermined timepoints during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented diagnosis of CD20+ Follicular lymphoma grade 1-2 or 3a, as defined in the 2017 edition of the World Health Organization (WHO) classification;
2. Age ≥ 18 years;
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (Appendix B);
4. No previous immunochemotherapy for the lymphoma (localized radiotherapy or rituximab monotherapy with max of 4 doses are allowed);
5. Ann Arbor stage II-IV (Appendix A);
6. High tumor burden as per Groupe d'Etude des Lymphomes Folliculaires (GELF) criteria defined as the presence of at least one of the following:

   * systemic symptoms;
   * Tumor bulk (any nodal or extranodal tumor mass with diameter > 7 cm);
   * involvement of ≥ 3 nodal sites, each with a diameter ≥ 3 cm;
   * splenomegaly;
   * compressive syndrome (organ compression);
   * serous effusion;
   * circulant malignant cells;
   * cytopenia;
   * Eastern Cooperative Oncology Group - Performance Status (ECOG-PS) > 1;
   * Lactate dehydrogenase (LDH) > upper limit of normality (ULN);
   * β2-microglobulin > 3 mg/L.
7. At least one site of measurable nodal disease at baseline ≥ 1.5 cm in the longest transverse diameter as determined by CT scan (MRI is allowed if CT scan cannot be performed); or evaluable disease at baseline FDG-PET (18F-fluorodeoxyglucose (FDG)-Positron Emission Tomography (PET)) scan (at least one metabolic active site of disease);
8. Adequate hematological counts (unless due to bone marrow involvement by lymphoma) defined as follows:

   1. Absolute Neutrophil count (ANC) > 1.5 x 109/L;
   2. Platelet count ≥ 80 x 109/L ;
   3. Hemoglobin ≥ 10 g/dL.
9. Adequate renal function defined as creatinine ≤ 2 mg/dL, unless secondary to lymphoma;
10. Adequate hepatic function defined as bilirubin ≤ 2 mg/dL, unless secondary to lymphoma;
11. Left Ventricular Ejection Fraction (LVEF) > 50% at bidimensional echocardiogram (mandatory only for patients receiving R/G-CHOP);
12. Life expectancy ≥ 6 months;
13. Subject understands and voluntarily signs an informed consent form approved by an Independent Ethics Committee (IEC) prior to the initiation of any screening or study-specific procedures;
14. Subject must be able to adhere to the study visit schedule and other protocol requirements;
15. Women of childbearing potential (WOCBP) and men must agree to use effective contraception if sexually active. This applies for the time period between signing of the informed consent form and 12 months after last rituximab dose or 18 months after last obinutuzumab dose. A woman is considered of childbearing potential, i.e. fertile, following menarche and until becoming postmenopausal unless permanently sterile. Permanent sterilization methods include but are not limited to hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for continuous 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. The investigator or a designated associate is requested to advise the patient how to achieve highly effective birth control (failure rate of less than 1%) e.g., intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner. The use of condoms by male patients is required (even if surgically sterilized, i.e., status post vasectomy) unless the female partner is permanently sterile. Full sexual abstinence is admitted when this is in line with the preferred and usual lifestyle of the subject, for the same time period planned for other methods of birth control (see above). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post ovulation methods for the female partner) and withdrawal are not acceptable methods of contraception).

Exclusion Criteria:

1. Histological diagnosis different from FL grade 1-3a WHO 2017 classification;
2. Suspect or clinical evidence of Central Nervous System (CNS) involvement by lymphoma;
3. Contraindication to the use of anti-CD20 monoclonal antibodies;
4. Subject has received any anticancer therapy (chemotherapy, immunotherapy, investigational therapy, including targeted small molecule agents) within 14 days prior to the first dose of study drug;
5. Noteworthy history of neurologic, psychiatric, endocrinological, metabolic, immunologic, or hepatic disease that would preclude participation in the study or compromise ability to give informed consent;
6. Any history of other active malignancies within 3 years prior to study entry, with the exception of: adequately treated in situ carcinoma of the cervix uterine; basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin; limited stage surgically removed breast cancer or adequately treated with radiation therapy; limited stage prostate carcinoma surgically removed or adequately treated with radiation therapy; previous malignancy confined and surgically resected with curative intent;
7. Evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

   * Uncontrolled and/or active systemic infection (viral, bacterial or fungal), including active ongoing infection from SARS-CoV-2;
   * Chronic or acute hepatitis B (HBV) or hepatitis C (HCV) requiring treatment. Note: subjects with serologic evidence of prior vaccination to HBV (i.e., HBsAg negative, HBsAb positive and HBcAb negative) or positive HBcAb from previous infection or intravenous immunoglobulins (IVIG) may participate; inactive carriers (HBsAg positive with undetectable HBV- DNA) are eligible. Patients with presence of HCV antibody are eligible only if Polymerase Chain Reaction (PCR) negative for HCV-RNA;
8. Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 605 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | The endpoint will be assessed from the beginning of the study up to 104 months (end of study)
  The length of time during and after the treatment that patients live with the disease, but it does not get worse. Progression-Free Survival (PFS) will be measured from the time of study entry to documented progression or to the patient's death as a result of any causes. Subjects with incomplete follow-up or with no disease evaluation will be censored at the date of last available documented status of freedom from failure.

SECONDARY OUTCOMES:
Overall Survival (OS) | The endpoint will be assessed from the beginning of the study up to 104 months (end of study)
  Overall Survival, the percentage of patients alive, will be measured from the time of study entry to death from any cause. Patients who have not died at the time of the final analysis will be censored at the date of the last contact.
Event-Free Survival (EFS) | The endpoint will be assessed from the beginning of the study up to 104 months (end of study)
  The measure of time after treatment that patients have not have cancer come back or get worse. It will be measured from the time of study entry to any treatment failure, including disease progression, or discontinuation of treatment for any reason (e.g., disease progression, toxicity, patient preference, initiation of a new treatment without documented progression) or death from any cause.
Overall Response rate (ORR) | The endpoint will be assessed from the beginning of the study up to 104 months (end of study)
  Overall response rate (ORR) is defined as the proportion of patients who have a partial or complete response to therapy; It will be defined according to Response Criteria for Non-Hodgkin Lymphoma (NHL) with Positron Emission Tomography (PET) (Lugano 2014). ORR will include the sum of patients in Complete Remission and Partial Remission (CR + PR). It will be evaluated on assessed patients and on all treated patients, considering patients without a response assessment (due to any reason) as non-responders.
  The best overall response will be defined as the best response between the date of beginning of therapy and the last restaging.
Complete response rate (CRR) | The endpoint will be assessed from the beginning of the study up to 104 months (end of study)
  The Complete Response Rate is defined as the percentage of patient in Complete Remission. It will be defined according to Response Criteria for Non-Hodgkin Lymphoma (NHL) with Positron Emission Tomography (PET) (Lugano 2014). CRR will include only patients in Complete Remission (CR). It will be evaluated on assessed patients and on all treated patients, considering patients without a response assessment (due to any reason) as non-responders.
Molecular response | The endpoint will be assessed from the beginning of the study up to 104 months (end of study)
  Molecular response assessed by means of the evaluation of the Bcl2/IgH rearrangement at baseline and of the Minimal Residual Disease (MRD) at subsequent defined timepoints.
Incidence of toxicities (Safety of the treatment) | The endpoint will be assessed from the beginning of the study up to 104 months (end of study)
  Safety of the treatment according to the current version of the CTCAE. Incidence of toxicities
Patient-Reported Outcomes (PROs) | The endpoint will be assessed from the beginning of the study up to 104 months (end of study)
  Health Related Quality of Life (HR-QoL) will be evaluated by means of Patient-Reported Outcome(s) PROs. Patients will be asked to complete the Functional Assessment of Cancer Therapy - Lymphoma (FACT-Lym) questionnaire at prespecified points during the study. The questionnaire results will be analyzed according to recommendations of the instrument scoring procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Luminari, MD, Principal Investigator — Reggio Emilia - Azienda Unitа Sanitaria Locale-IRCCS - Arcispedale Santa Maria Nuova - Ematologia
Locations (71):
- Italy (71):
  - Ospedale "Monsignor Raffaele Dimiccoli" - Ematologia, Barletta, Barletta Andria Trani
  - Casa Sollievo della Sofferenza - U.O. Ematologia, San Giovanni Rotondo, Foggia
  - IRCCS Istituto Romagnolo per lo studio dei Tumori "Dino Amadori" - IRST S.R.L. - Ematologia, Meldola, Forlì - Cesena
  - A.O. C. Panico - U.O.C Ematologia e Trapianto, Tricase, Lecce
  - Nuovo Ospedale Civile di Sassuolo - Day Hospital Oncologico, Sassuolo, Modena
  - ASST MONZA Ospedale S. Gerardo - Ematologia, Monza, Monza E Brianza
  - IRCCS Centro di Riferimento Oncologico di Aviano - Divisione di Oncologia e dei Tumori immuto-correlati, Aviano, Pordenone
  - Presidio ospedaliero "A. TORTORA" - U.O. Onco-ematologia, Pagani, Salerno
  - Fondazione del Piemonte per l'Oncologia - IRCCS - Ematologia, Candiolo, Torino
  - Ospedale di Castelfranco Veneto - Ematologia, Castelfranco Veneto, Treviso
  - ASST Valle Olona - Ospedale di Circolo di Busto Arsizio - S.C. Ematologia, Busto Arsizio, Varese
  - Ospedale Dell'Angelo - U.O. Ematologia, Mestre, Venezia
  - USLL13 - Dipartimento di Scienze Mediche UOC di Oncologia ed Ematologia Oncologica, Mirano, Venezia
  - A.O. SS. Antonio e Biagio e Cesare Arrigo - S.C. Ematologia, Alessandria
  - AOU Ospedali Riuniti - Clinica di Ematologia, Ancona
  - Ospedale C.e G. Mazzoni - U.O.C. di Ematologia, Ascoli Piceno
  - Azienda Ospedaliera S.Giuseppe Moscati - S.C. Ematologia e Trapianto emopoietico, Avellino
  - AOU Policlinico Consorziale - U.O. Ematologia con Trapianto, Bari
  - IRCCS Istituto Tumori Giovanni Paolo II - U.O.C Ematologia, Bari
  - Ospedale S. Martino - UOC Oncologia, Belluno
  - A.O.R.N. Gaetano Rummo - DH Ematologico, Benevento
  - Nuovo Ospedale degli Infermi - SSD Ematologia, Biella
  - ASST Spedali Civili di Brescia - Ematologia, Brescia
  - Ospedale Antonio Perrino - U.O. Ematologia e Trapianti di Midollo, Brindisi
  - Azienda Ospedaliero - Universitaria Policlinico - Vittorio Emanuele Presidio Ospedale Ferrarotto - Ematologia, Catania
  - AO Pugliese Ciaccio - SOC Ematologia, Catanzaro
  - Azienda Ospedaliera di Cosenza - UOC Ematologia, Cosenza
  - A.O. S. Croce e Carle - S.C. di Ematologia e Trapianto di Midollo Osseo, Cuneo
  - Azienda Ospedaliero-Universitaria di Ferrara - Arcispedale Sant'Anna - Ematologia e fisiopatologia della coagulazione, Ferrara
  - Azienda Ospedaliera Universitaria Careggi - Unitа funzionale di Ematologia, Florence
  - Ospedale San Giovanni di Dio - SOS Ematologia clinica e oncoematologia ASL Toscana Centro, Florence
  - Ospedale Policlinico San Martino S.S.R.L. - IRCCS per l Oncologia - Ematologia, Genova
  - Ospedale Vito Fazzi - Ematologia, Lecce
  - Azienda Ospedali Riuniti Papardo-Piemonte - S.C. Ematologia, Messina
  - Istituto Scientifico San Raffaele - Unitа Linfomi - Dipartimento Oncoematologia, Milan
  - ASST Santi Paolo e Carlo - Onco - Ematologia, Milan
  - ASST Grande Ospedale Metropolitano Niguarda - SC Ematologia, Milan
  - Ospedale Maggiore Policlinico - Fondazione IRCCS Ca Granda - Ematologia, Milan
  - AOU Universitа degli Studi della Campania Luigi Vanvitelli - Oncologia Medica ed Ematologia, Napoli
  - AOU Maggiore della Caritа di Novara - SCDU Ematologia, Novara
  - I.R.C.C.S. Istituto Oncologico Veneto - Oncologia 1, Padua
  - AOU di Padova - Ematologia, Padua
  - AOU Policlinico Giaccone - Ematologia, Palermo
  - A.O. Ospedali Riuniti Villa Sofia-Cervello - Divisione di Ematologia, Palermo
  - UO Ematologia e CTMO - AOU di Parma, Parma
  - IRCCS Policlinico S. Matteo di Pavia - Div. di Ematologia, Pavia
  - P.O. Spirito Santo di Pescara - UOS Dipartimentale - Centro di diagnosi e Terapia dei linfomi, Pescara
  - Ospedale Guglielmo da Saliceto - U.O.Ematologia, Piacenza
  - AOU Pisana - U.O. Ematologia, Pisa
  - A.O.R. "San Carlo" - U.O. Ematologia, Potenza
  - Ospedale S. Stefano - SOS Oncoematologia, ASL Toscana Centro, Prato
  - Ospedale delle Croci - Ematologia, Ravenna
  - Grande Ospedale Metropolitano Bianchi Melacrino Morelli - Ematologia, Reggio Calabria
  - Azienda Unitа Sanitaria Locale-IRCCS - Arcispedale Santa Maria Nuova - Ematologia, Reggio Emilia
  - Ospedale degli Infermi di Rimini - U.O. di Ematologia, Rimini
  - Policlinico Tor Vergata - Ematologia, Roma
  - Ospedale S. Eugenio - UOC Ematologia, Roma
  - Ospedale S. Camillo - Ematologia, Roma
  - Policlinico Umberto I - Universitа "La Sapienza" - Istituto Ematologia -Dipartimento di Medicina Traslazionale e di Precisione, Roma
  - Universitа Cattolica S. Cuore - Ematologia, Roma
  - Ospedale di Rovigo - S.O.S. Oncoematologia, Rovigo
  - Ematologia e Trapianti A.O. San Giovanni di Dio e Ruggi D Aragona - U.O. Ematologia, Salerno
  - AOU di Sassari - Ematologia, Sassari
  - AOU Senese - U.O.C. Ematologia, Siena
  - Azienda Ospedaliera della Valtellina e della Valchiavenna P.O. Sondrio - Medicina Interna - Centro Malattie del Sangue P.O. Sondrio, Sondrio
  - A.O. S. Maria di Terni - S.C. Oncoematologia, Terni
  - A.O.U. Citta della Salute e della Scienza di Torino - Ematologia Universitaria, Torino
  - A.O.U. Citta della Salute e della Scienza di Torino - S.C.Ematologia, Torino
  - San Giovanni Bosco - ASL Cittа di Torino - SSD di Ematologia e Malattie Trombotiche, Torino
  - Ospedale Ca Foncello - S.C di Ematologia, Treviso
  - Azienda Sanitaria Universitaria Giuliano Isontina (ASUGI) - SC Ematologia, Trieste

IPD SHARING:
Plan to Share IPD: No